CLINICAL TRIAL: NCT04603261
Title: Time to Excretion of Contrast, a Maastricht Prospective Observational Study
Acronym: TEMPOS
Status: Withdrawn | Type: Observational
Why Stopped: delayed
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL.MUMC.AMACINGrp.2
Record Dates: First submitted 2020-10-07; First posted 2020-10-26 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Renal Insufficiency; Acute Kidney Injury; Contrast-induced Nephropathy
Keywords: intravascular iodinated contrast; contrast-induced acute kidney injury; post-contrast acute kidney injury; iodinated contrast elimination time; contrast retention; delayed contrast elimination
MeSH Terms: conditions — Renal Insufficiency; Acute Kidney Injury | interventions — Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and urine samples may be stored for renal injury biomarker assays
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- eGFR <30 mL/min/1.73m2: Patients with eGFR <30 mL/min/1.73m2 in absence of dialysis referred for an elective procedure with intravascular administration of iodinated contrast material at Maastricht UMC+.
  Interventions: Diagnostic Test: Contrast concentration in urine
- eGFR 30-59 mL/min/1.73m2: For each included patient with eGFR <30 mL/min/1.73m2, two patients matched for age, sex and contrast procedure type will be included: one with eGFR 30-59 mL/min/1.73m2 and one with eGFR >=60 mL/min/1.73m2.
  Interventions: Diagnostic Test: Contrast concentration in urine
- eGFR >=60 mL/min/1.73m2: For each included patient with eGFR <30 mL/min/1.73m2, two patients matched for age, sex and contrast procedure type will be included: one with eGFR 30-59 mL/min/1.73m2 and one with eGFR >=60 mL/min/1.73m2.
  Interventions: Diagnostic Test: Contrast concentration in urine

INTERVENTIONS:
Diagnostic Test: Contrast concentration in urine — Iodinated contrast content of urine samples, collected post-contrast over a period of 5 days at all times of natural excretion within that period, will be assayed.
  Serum creatinine will be measured daily before (day 0) and during 5 days post-contrast, and again at 1 month post-contrast.

SUMMARY:
Risk of contrast-induced kidney injury is expected to be strongly correlated with exposure time. Studies on the excretion of iodinated contrast material are few and have mostly been carried out in patients with normal renal function. Although case wise reports of persistent renograms have been published, it is not known how long contrast is retained before excretion in patients with eGFR <30 mL/min/1.73m2, nor which of these patients are most susceptible to contrast retention. The current observational study aims to compare contrast elimination time and % contrast excretion in patients with eGFR <30 mL/min/1.73m2, to matched patients (for age, sex and contrast procedure type) with eGFR 30-59 and eGFR >=60 mL/min/1.73m2.

DETAILED DESCRIPTION:
The primary aim of the current study is to determine contrast elimination time and % in three groups of patients, (with severely reduced, moderate, and mildly reduced to normal renal function). Secondary aims are to explore whether specific situations/characteristics result in higher probability of delayed elimination of contrast, and whether there is a link between elimination time and adverse post-contrast outcomes (post-contrast incidences of acute kidney injury; post-contrast changes in eGFR within 5 days from baseline; 1-month post-contrast change in eGFR; 1-month post-contrast incidences of eGFR decline >=5 mL/min/1.73m2; 1-month dialysis and mortality).

ELIGIBILITY:
Inclusion Criteria:

- eGFR <30 mL/min/1.73m2 in absence of dialysis referred for an elective procedure with intravascular administration of iodinated contrast material at Maastricht UMC+

For each included patient with eGFR <30 mL/min/1.73m2, two matched patients will be included:

* 1. eGFR 30-59 mL/min/1.73m2 referred for an elective procedure with intravascular administration of iodinated contrast material at Maastricht UMC+ with age, sex and contrast procedure type matching the age, sex and contrast procedure type of an eGFR <30 mL/min/1.73m2 participant.
* 2. eGFR >=60 mL/min/1.73m2 referred for an elective procedure with intravascular administration of iodinated contrast material at Maastricht UMC+ with age, sex and contrast procedure type matching the age, sex and contrast procedure type of an eGFR <30 mL/min/1.73m2 participant.

Exclusion Criteria:

* age <18 years
* dialysis or pre-dialysis
* intravascular contrast administration having occurred <30 days before the first baseline sample
* emergency or intensive care status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive eligible patients with eGFR <30 mL/min/1.73m2 and matched eGFR 30-59 mL/min/1.73m2 and eGFR >=60 mL/min/1.73m2 patients referred for an elective procedure with intravascular iodinated contrast at Maastricht UMC+
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2097-11-01 (Estimated); Primary Completion 2099-11-01 (Estimated); Study Completion 2099-11-01 (Estimated)

PRIMARY OUTCOMES:
time to contrast-free urine. | 5 days
  time to the first contrast-free urine sample from the time of intravascular iodinated contrast administration. Time to contrast-free urine will be compared between three groups of patients (with eGFR <30 mL/min/1.73m2, eGFR 30-59 mL/min/1.73m2, and eGFR >=60 mL/min/1.73m2).

SECONDARY OUTCOMES:
% contrast elimination. | 5 days
  percentage of total contrast administered excreted in urine within 5 days. Percentage contrast elimination will be compared between three groups of patients (with eGFR <30 mL/min/1.73m2, eGFR 30-59 mL/min/1.73m2, and eGFR >=60 mL/min/1.73m2).
contrast elimination versus adverse post-contrast outcomes. | 1 month
  The underlying hypothesis is that delayed elimination increases contrast toxicity which increases adverse event risk. This will be explored by comparing percentages with post-contrast adverse events (acute kidney injury; changes in eGFR; eGFR decline ≥5mL/min/1.73m2; dialysis; mortality; up to 1-month) in groups with and without delayed elimination, stratified by eGFR (<30, 30-59, ≥60). Relevant patient and procedural characteristics will also be compared to identify potential predictors of delayed elimination.
  Contrast elimination times are unknown, therefore 'delayed' is defined as time to contrast-free urine exceeding patient group median value. In clinical practice, normal contrast elimination is assumed to be ≥24h. Therefore, 1. Normal (≤24h); 2. Delayed (24-48h); 3. Severely delayed (>48h) elimination subgroups will also be compared. Subgroup cut-off values may be added at a later stage (e.g., in the event of many or no patients with elimination >48h).

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht UMC, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No